CLINICAL TRIAL: NCT02593006
Title: Start Time Optimization of Biologics in Polyarticular JIA
Acronym: STOP-JIA
Status: Completed | Type: Observational
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Childhood Arthritis and Rheumatology Research Alliance (Other); Duke Clinical Research Institute (Other); Seattle Children's Hospital (Other); Children's Hospital of Philadelphia (Other); Boston Children's Hospital (Other); The Hospital for Sick Children (Other); University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: Pro5835
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Results first posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Polyarticular Juvenile Rheumatoid Arthritis; Arthritis, Juvenile Idiopathic
Keywords: Joint Diseases; Juvenile Arthritis; treatment; biologic therapy; comparative effectiveness
MeSH Terms: conditions — Arthritis, Juvenile; Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
STOP-JIA is a PCORI funded prospective observational study which compared the clinical effectiveness and impact on patient reported outcomes of 3 Childhood Arthritis & Rheumatology Research Alliance (CARRA) consensus derived treatment strategies (CTPs) in new-onset polyarticular JIA (pJIA) patients to answer the critical question of when is the best time to begin biologic medications to achieve the optimal clinical and patient reported outcomes. Because the CARRA Registry will be used for data collection, all patients will be enrolled in the CARRA Registry. The standard of care treatments are chosen by the treating physician and patient/caregiver and are not randomized.

DETAILED DESCRIPTION:
STOP-JIA is a prospective, observational study comparing the clinical effectiveness and impact on patient reported outcomes of 3 different treatment strategies (CTPs) in new onset pJIA patients to answer the critical question of when to start biologic medications. All participants will be enrolled in the CARRA Registry and started on one of the CTPs, which will be decided by the treating physician and patient/caregiver. Subjects will be enrolled at one of 60 participating CARRA sites across the US and Canada. Total anticipated enrollment was 400 and this was completed in 9/19.

Specific Aim 1:

To compare the clinical effectiveness of different strategies (CTPs) for using biologic medications in achieving clinically inactive disease (CID) at 12 months in new-onset pJIA. Three common strategies that differ in the timing of biologic medication introduction will be compared: 1) Step-Up: disease modifying anti-rheumatic drug (DMARD) monotherapy stepping up by addition of a biologic medication if needed; 2) Early Combination: DMARD plus biologic medication at treatment onset; and 3) Biologic First: biologic medication monotherapy at treatment onset.

Hypothesis 1: A significantly higher proportion of children started on a biologic medication at onset (CTP 2 or 3) will achieve CID after 12 months of therapy compared to standard therapy (CTP 1).

Specific Aim 2:

To compare patient and caregiver reported outcomes between the different strategies.

Hypothesis 2: There will be statistically significant differences in patient/caregiver reported outcomes (PROs) between treatment strategies that can inform future patients and providers in selecting optimal treatments.

The CARRA Registry will be housed at CARRA's clinical and data coordinating center, Duke Clinical Research Institute (DCRI). The CARRA Registry Protocol documents that the CARRA Registry fulfills all PCOR standards for registries. STOP-JIA will utilize data collection, storage, and management processes, systems requirements, and security processes already established for the CARRA Registry at DCRI.

STOP-JIA used Web-based electronic CRFs (eCRFs) developed for the CARRA Registry that are already familiar to site personnel. The eCRF platform, RAVE, is 21CFR part11 compliant and meets regulatory requirements. Database and Web servers are secured by a firewall and through controlled physical access. eCRFs will be monitored for completeness, accuracy, and attention to detail throughout the study by DCRI data and site management teams using processes developed for the CARRA Registry and consistent with DCRI's internal SOPs. Use of electronic data capture will allow for immediate prompts/queries if entered values are out of expected ranges or there are incomplete data fields. The design of the data collection instrument will allow centers to record a planned assessment of a patient was missed and to enter any known reasons for the assessment being missed. DCRI will regularly provide reports detailing data completion metrics to the sites. Stakeholder engagement is also an important aspect of this study, and patients/caregivers as well as other stakeholders are serving as research partners and advisors in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age less than 19 at baseline (if 18 or older, agrees to be followed for at least one year)
* Diagnosis of Arthritis per ACR definition.
* Arthritis present in one joint for a least six weeks
* At least 5 active joints at baseline
* Contraception if sexually active (male and female)

May have any of the following:

* RF+ polyarticular JIA
* RF- polyarticular JIA
* Extended oligoarticular JIA
* Psoriatic JIA
* Enthesitis related JIA
* Undifferentiated JIA
* Psoriasis
* Sacroiliitis
* Uveitis
* Enthesitis
* Prior treatments permitted:

  * NSAIDS
  * Hydroxychloroquine
  * Intraocular / topical / intraarticular glucocorticoids
  * IV or PO steroids if one of the below criteria are met:

    --If treated ≤ 3 months prior to baseline: treatment cannot exceed 2 weeks

    --If treated > 3 months prior to baseline: any treatment course is permitted as long as treatment was completed 90 days prior to baseline
  * Methotrexate started no more than 1 month prior to the baseline visit
  * Biologics - received only 1 dose within 1 week of the baseline visit

Exclusion Criteria:

* Features consistent with systemic JIA
* Treatment with any medications for JIA aside from those listed above.
* Known inflammatory bowel disease
* Known celiac disease
* Known Trisomy 21
* History of or current malignancy
* Concomitant serious active or recurrent chronic bacterial, fungal or viral infection
* Significant organ system disorder limiting use of treatments for pJIA
* Live vaccine within a month prior to baseline

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with new onset, untreated Poly JIA enrolled in the CARRA Registry.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2015-11; Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yukiko Kimura, MD, Principal Investigator — Hackensack Meridian Health; Sarah Ringold, MD, Principal Investigator — Seattle Children's Hospital
Locations (55):
- United States (52):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University Medical Center, Palo Alto, California
  - Rady Children's Hospital-San Diego, San Diego, California
  - University of California at San Francisco Medical Center, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - University of Florida Shand's Children's Hospital, Gainesville, Florida
  - Emory Children's Center, Atlanta, Georgia
  - Georgia Regents University Medical Center, Augusta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville School of Medicine, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Baystate Medical Center, High Street Health Center, Springfield, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Saint Louis University School of Medicine, St Louis, Missouri
  - Saint Louis Children's Hospital, St Louis, Missouri
  - HackensackUniversity Medical Center, Hackensack, New Jersey
  - Goryeb Children's Hospital, Morristown, New Jersey
  - Pediatric Specialty Center at Saint Barnabas, West Orange, New Jersey
  - Albany Medical College, Albany, New York
  - Cohen Children's Medical Center of New York, Lake Success, New York
  - New York University Langone Medical Center, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Columbia University Medical Center, New York, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Levine Children's Hospital, Charlotte, North Carolina
  - Duke Children's Hospital & Health Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - UH Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Clevland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Randall Children's Hospital at Legacy Emanuel, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina Children's Hospital, Charleston, South Carolina
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - University of Texas Southwestern Medical Center Dallas, Dallas, Texas
  - Baylor College of Medicine Pediatric Immunology, Allergy and Rheumatology, Houston, Texas
  - University of Utah Hospitals and Clinics, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin-American Family Children's Hospital, Madison, Wisconsin
- Canada (3):
  - University of Calgary- Alberta Children's Hospital, Calgary, Alberta
  - IWK Health Center, Halifax, Nova Scotia
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Key outcome data, treatment data and baseline characteristics will be shared with other researchers upon request and are subject to the CARRA data and sample sharing policy (https://carragroup.org/UserFiles/file/CARRA-DATA-SAMPLE-SHARING-POLICY-04November2016.pdf). Documentation of appropriate IRB/ethics board approval will be required.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be available for requests through the CARRA data and sample request portal once the PCORI Final Research Report has been approved and is publicly available. There is no time limit.
Access Criteria: Investigators may request data through the CARRA data and sample share request portal. Inquiries may be sent to research@carragroup.org.

REFERENCES:
- [Derived] Kimura Y, Schanberg LE, Tomlinson GA, Riordan ME, Dennos AC, Del Gaizo V, Murphy KL, Weiss PF, Natter MD, Feldman BM, Ringold S; CARRA STOP-JIA Investigators. Optimizing the Start Time of Biologics in Polyarticular Juvenile Idiopathic Arthritis: A Comparative Effectiveness Study of Childhood Arthritis and Rheumatology Research Alliance Consensus Treatment Plans. Arthritis Rheumatol. 2021 Oct;73(10):1898-1909. doi: 10.1002/art.41888. Epub 2021 Sep 3. PMID 34105312
- [Derived] Ong MS, Ringold S, Kimura Y, Schanberg LE, Tomlinson GA, Natter MD; CARRA Registry Investigators. Improved Disease Course Associated With Early Initiation of Biologics in Polyarticular Juvenile Idiopathic Arthritis: Trajectory Analysis of a Childhood Arthritis and Rheumatology Research Alliance Consensus Treatment Plans Study. Arthritis Rheumatol. 2021 Oct;73(10):1910-1920. doi: 10.1002/art.41892. Epub 2021 Aug 27. PMID 34105303
- See also: Click here for more information on the Observational Study of Pediatric Rheumatic Diseases: The CARRA Registry — https://www.clinicaltrials.gov/ct2/show/NCT02418442?term=carra&rank=2

RESULTS

PARTICIPANT FLOW:
Groups:
- Step-Up CTP: Consensus Treatment Plan where subjects begin non biologic DMARD (methotrexate, sulfasalazine, or leflunomide) stepping up to biologic if not improved by 3 months
- Early Combination CTP: Consensus Treatment Plan where patients start a DMARD(methotrexate, sulfasalazine, or leflunomide) and biologic treatment within one month of each other.
- Biologic Frist CTP: Consensus Treatment Plan where patients begin Biologic treatment
Period: Overall Study
Arm/Group | Step-Up CTP | Early Combination CTP | Biologic Frist CTP
Started | 257 | 100 | 43
Completed | 250 | 93 | 38
Not Completed | 7 | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Step-Up CTP | Early Combination CTP | Biologic Frist CTP | Total
Number analyzed (Participants) | 257 | 100 | 43 | 400
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 257 | 99 | 43 | 399
  Between 18 and 65 years | 0 | 1 | 0 | 1
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 11.07 [1.10 to 17.85] | 11.38 [1.15 to 18.41] | 12.34 [1.40 to 17.95] | 11.28 [1.10 to 18.41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 192 | 75 | 27 | 294
  Male | 65 | 25 | 16 | 106
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 0 | 3
  Asian | 15 | 4 | 2 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 15 | 5 | 3 | 23
  White | 188 | 68 | 27 | 283
  More than one race | 9 | 3 | 5 | 17
  Unknown or Not Reported | 27 | 19 | 6 | 52
Region of Enrollment [Number; unit: participants]
  Canada | 32 | 2 | 1 | 35
  United States | 225 | 98 | 42 | 365
Clinical Juvenile Arthritis Disease Activity Score [Mean (Standard Deviation); unit: units on a scale] — The cJADAS-10 is a clinical measure of disease activity that is a sum of the active joint count (up to 10), physician global assessment of disease activity measured on a 0 to 10 visual analog scale where 0=no activity and 10 =maximum activity; patient/parent rating of well-being assessed on a 0 to 10 visual analog scale where 0=very well and 10= very poor; cJADAS-10 Score range is 0-30, where composite score < or = 2.5 - low disease activity; 2.51-8.5 -Moderate disease activity, > 8.5- High disease activity.
  units on a scale | 17.08 (4.55) | 20.18 (4.37) | 19.05 (4.29) | 18.08 (4.67)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinically Inactive Disease (CID) Off Glucocorticoids
Description: This is a provisional criteria which describes a state of complete disease inactivity in Juvenile Idiopathic Arthritis (JIA). We will assess the proportion of patients achieving CID off glucocorticoids in each treatment arm.
Time Frame: 12 months after baseline
Population: Subjects are children and adolescents between the ages of 2 and 18 who are newly diagnosed with a polyarticular form of JIA and treated for 12 months with one of the consensus treatment plans.
  328 participants had complete data for the primary CID endpoint at 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants achieving CID
Groups:
- Step-Up Consensus Treatment Plan (CTP): Initial therapy with a non biologic Disease Modifying Anti-Rheumatic Drug (DMARD) stepping up to a biologic treatment if needed
- Early Combination CTP: Initial therapy with a non-biologic DMARD and biologic treatment at the start of treatment
- Biologic First CTP: Initial therapy with a biologic treatment without a non-biologic DMARD
Arm/Group | Step-Up Consensus Treatment Plan (CTP) | Early Combination CTP | Biologic First CTP
Number analyzed (Participants) | 217 | 78 | 33
percentage of participants achieving CID | 32.3 [26.2 to 39.0] | 37.2 [26.7 to 48.9] | 24.2 [11.7 to 42.6]
Statistical Analysis 1: Comparison: Step-Up Consensus Treatment Plan (CTP) vs Early Combination CTP vs Biologic First CTP; Test type: Superiority; p > 0.05, Propensity weighted regression model; Risk Difference (RD) = 10.3, 95% CI 2-sided [-3.2 to 23.8]

2. Secondary Outcome: Comparison of PROMIS Pain and Mobility Scores Between the 3 Consensus Treatment Plan Groups
Description: The Patient Reported Outcomes Measurement Information System (PROMIS) pain interference and mobility scores will be compared between the 3 CTP groups. Pain interference scores range from 0-100 and higher scores are worse. Mobility scores also range from 0-100 and higher scores are better.
Time Frame: 12 months after baseline
Population: Same description as above for the population for the primary outcome
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Step-Up CTP: Initial therapy with a non biologic Disease Modifying Anti-Rheumatic Drug (DMARD) stepping up to a biologic treatment if needed
Arm/Group | Step-Up CTP | Early Combination CTP | Biologic First CTP
Number analyzed (Participants) | 257 | 100 | 43
score on a scale
  Pain Interference: number analyzed (Participants) | 188 | 75 | 35
  Pain Interference | 53.1 (10.0) | 55.5 (9.2) | 55.9 (9.3)
  Mobility: number analyzed (Participants) | 195 | 74 | 35
  Mobility | 38.6 (10.3) | 35.8 (9.1) | 37.5 (9.1)
Statistical Analysis 1: Comparison: Step-Up CTP vs Early Combination CTP vs Biologic First CTP; Test type: Superiority; p = 0.04, Mixed Models Analysis — Global test of interaction between time and treatment group

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Baseline through Study completion. For each participant, the time period was on average 1 year
Arm/Group | Step-Up CTP | Early Combination CTP | Biologic First CTP
All-Cause Mortality (participants affected / at risk) | 0/257 | 0/100 | 0/43
Serious Adverse Events (participants affected / at risk) | 12/257 | 3/100 | 5/43
Other Adverse Events (participants affected / at risk) | 19/257 | 5/100 | 1/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Step-Up CTP (N=257) | Early Combination CTP (N=100) | Biologic First CTP (N=43)
Hip Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Cervical Spine Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Compund Fracture Ulna & Radius (Injury, poisoning and procedural complications) | 0 | 1 | 0
Depression with Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 1
Influenza (General disorders) | 2 | 0 | 0
Infections treated with IV antibiotics (Infections and infestations) | 2 | 1 | 2
Inflammatory Bowel Disease (Gastrointestinal disorders) | 1 | 0 | 0
Drug induced Lupus (Immune system disorders) | 1 | 0 | 0
hip effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Shingles (Infections and infestations) | 0 | 0 | 1
Vertigo (Nervous system disorders) | 0 | 0 | 1
Worsening Bipolar Affective Disorder (Psychiatric disorders) | 1 | 0 | 0
Macrophage Activation Syndrome (Immune system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Step-Up CTP (N=257) | Early Combination CTP (N=100) | Biologic First CTP (N=43)
Hepatitis (Hepatobiliary disorders) | 3 | 2 | 0
Hypersensitivity Reaction (Immune system disorders) | 1 | 0 | 0
Inflammatory Bowel Disease (Gastrointestinal disorders) | 1 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Uveitis (New Onset) (Eye disorders) | 9 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT02593006/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT02593006/SAP_001.pdf